CLINICAL TRIAL: NCT03643081
Title: Evaluation of the Interest of the Medical Device Called "Fluobeam" in the Localization, Visualization of the Parathyroid Glands for Patients With Mild Primary Hyperparathyroidism. A Randomized Controled Prospective Open -Labeled Monocentric Study.
Brief Title: Evaluation of the Interest of the Medical Device Called "Fluobeam" in the Localization, Visualization of the Parathyroid Glands for Patients With Mild Primary Hyperparathyroidism
Acronym: FLUO-PARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC18_0260
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Mild Primary Hyperparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- use of camera "Fluobeam" (Experimental)
  Interventions: Device: Use of the camera "Fluobeam"
- Without use of the camera "Fluobeam" (No Intervention)

INTERVENTIONS:
Device: Use of the camera "Fluobeam" — Use of the camera "Fluobeam" to localize, visualize the parathyroid glands during a parathyroidectomy.
  Arms: use of camera "Fluobeam"

SUMMARY:
The aim of our study is to evaluate the value of the camera called "Fluobeam" in the localization, visualization of the parathyroid glands for patients with mild primary hyperparathyroidism.

DETAILED DESCRIPTION:
Recently, it has been shown that parathyroid glands presented auto fluorescence, visible in the near infra-red light. Parathyroid glands emit at 822 nanometers when they are stimulated by a laser of 785 nanometers. Fluoptics Company (Fluoptics SAS, Grenoble, France) will provide a camera called "Fluobeam", facilitating the visualization of the parathyroid glands. The fluorescence intensity of the parathyroid glands is much more elevated than that of the surrounding tissues.

Preliminary work showed the interest of this technique. Benmiloud and collabortors have shown that the utilization of the "Fluobeam" enable to decrease the post total thyroidectomy hypocalcemia rate by a better visualization and preservation of the parathyroid glands.

The aim of this study is to evaluate the value of "Fluobeam" in the localization, visualization of the parathyroid glands for patients with mild primary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 80 years old.
* Given signed written informed consent.
* Patient with moderated and sporadic primary hyperparathyroism (albumin-corrected serum calcium ≤2.85 mmol/l) requiring to be operated on.
* Patient affiliated to a social security system.

Exclusion Criteria:

* Underage and adults under guardianship.
* Pregnant or breast feeding women.
* Patients with history of cervical radiotherapy or cervicotomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
To compare the time required for the parathyroidectomy with or without the utilization of the camera "Fluobeam". | At Day 1(parathyroidectomy)

SECONDARY OUTCOMES:
To compare the results of the parathyroidectomy with or without the utilization of the camera "Fluobeam" in term of biological recovery. | At 6 months post parathyroïdectomy
  To compare the results of the parathyroidectomy with or without the utilization of the camera "Fluobeam" in term of biological recovery determined by normocalcemia (2,20 mmol/L < calcium < 2,60 mmol/L) at 6 months post surgery.
To compare the results of the surgery with or without the utilization of the "Fluobeam" in term of number of visualized parathyroid glands. | At Day 1(parathyroidectomy)
To compare the results of the surgery with or without the utilization of the "Fluobeam" in term of post-surgery laryngeal paralysis. | At 6 months post parathyroïdectomy
To compare the results of the surgery with or without the utilization of the "Fluobeam" in term of parathyroid morbidity (hypocalcemia with calcémia below 2 mmol/L) | At 6 months post parathyroïdectomy
To compare the results of the surgery with or without the utilization of the "Fluobeam" in term of cost-utility analysis according to the societal perspective and over a 6 months' time horizon of the surgery. | At 6 months post parathyroïdectomy

CONTACTS AND LOCATIONS:
Overall Officials: Eric MIRALLIE, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No